CLINICAL TRIAL: NCT04869306
Title: Effect of Hyaluronic Acid on Early and Late Tissue Healing After Removal of Impacted Mandibular Third Molars - A Double-blind, Randomized Controlled Clinical Trial
Brief Title: Effect of Hyaluronic Acid on Tissue Healing After Removal of Impacted Mandibular Third Molars (LM3)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Danijel Domic DMD, Dental medical doctor, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2244/2020
Record Dates: First submitted 2021-04-16; First posted 2021-05-03 (Actual); Last update posted 2022-09-01 (Actual); Status verified 2022-08

CONDITIONS: Tooth, Impacted
MeSH Terms: conditions — Tooth, Impacted

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Hyaluronic acid (Active Comparator): hyaluronic acid gel application after lower third molar removal
  Interventions: Device: Hyaluronic acid gel
- Hyaluronic acid+carrier (Active Comparator): hyaluronic acid gel application together with a carrier after lower third molar removal
  Interventions: Device: Hyaluronic acid gel + carrier
- Standard treatment (No Intervention): standard treatment after lower third molar removal (i.e., blood clot only)

INTERVENTIONS:
Device: Hyaluronic acid gel — After lower third molar removal, the test group 1 will additionally receive hyaluronic acid gel prior to wound closure.
  Arms: Hyaluronic acid
Device: Hyaluronic acid gel + carrier — After lower third molar removal, the test group 2 will additionally receive hyaluronic acid gel with a collagen carrier prior to wound closure.
  Arms: Hyaluronic acid+carrier

SUMMARY:
Hyaluronic acid (HY) is used in dentistry to improve wound healing after oral and periodontal surgical interventions. After the application of HY, a positive effect on the wound healing of extraction sockets and periodontal defects has been described. The removal of a mandibular wisdom tooth (LM3) often leads to remaining residual defects with increased probing depths distal to the second molar. To date, the influence of HY on periodontal healing of the distal aspect of the second molar after removal of the LM3 has not yet been investigated. Accordingly, the aim of this double-blind, controlled and randomized clinical study is the influence of the application of HY Gel or HY Gel in combination with an absorbable collagen sponge on the periodontal healing of the second molar after surgical removal of the LM3 compared to the standard procedure (blood clot). A total of 102 patients with an impacted LM3 and a pre-existing bone defect of at least 5 mm distal to the second molar will be included. In the HY test group (n = 34), HY gel is applied to the LM3 extraction socket, and in the HY + C test group (n = 34) HY gel and an absorbable collagen sponge, while the control group (n = 34) does not receive any additional treatment. Patients are followed up for 12 months and the presence of an increased probing depth (≥ 5mm) on the distal side of the second molar is defined as the main parameter. A more stable blood clot and thus improved wound healing including periodontal healing is expected through the use of HY.

ELIGIBILITY:
Inclusion Criteria:

1. Patients elder than 18 years;
2. uni- or bilateral vertical or mesioangular complete impaction of the LM3 classified to:
3. group II- or III- B or C according to Pell-Gregory (1933);
4. a distance ≥ 5 mm from the CEJ to marginal bone level at the distal aspect of the second molar.

Exclusion Criteria:

1. Patients with chronic diseases and/or
2. taking any medication, influencing hard and soft tissue healing;
3. acute pain/infection of the surgical region;
4. untreated periodontal disease;
5. patients smoking > 10 cigarettes per day;
6. pregnancy;
7. history of hypersensitivity or allergy to HY;
8. absence of an adjacent second molar;
9. presence of caries or restoration on the distal aspect of the adjacent second molar; and
10. inability to attend the follow-up appointments.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2021-11-29 (Actual); Primary Completion 2023-05-01 (Estimated); Study Completion 2023-05-01 (Estimated)

PRIMARY OUTCOMES:
Probing depth at adjacent second molar | 1 year
  Probing depth will be measured from the gingival margin to the bottom of the periodontal pocket measured in mm with a graduated periodontal probe at disco-buccal, distal and disco-lingual aspect of the second molar

CONTACTS AND LOCATIONS:
Locations (1):
- University Clinic of Dentistry, Medical University of Vienna, Vienna, Austria